CLINICAL TRIAL: NCT00429702
Title: Phase II Randomized, Double-Blinded Study of an Antiemetic Pump, Using Benadryl®, Avitan® and Decadron® (BAD), for Children Receiving Moderately or Highly Emetogenic Chemotherapy
Brief Title: Diphenhydramine, Lorazepam, and Dexamethasone in Treating Nausea and Vomiting Caused By Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to poor accrual and lack of feasibility to finish study per DSMB
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SCUSF 0503; SCUSF-0503 (Other: SunCoast CCOP Research Base); HLMCC-0503 (Other: H. Lee Moffitt Cancer Center Research Base); U10CA081920 (NIH)
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Results first posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-06

CONDITIONS: Nausea; Vomiting; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: nausea; vomiting; emetic chemotherapy; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Nausea; Vomiting | interventions — Calcium Dobesilate; Dexamethasone; Diphenhydramine; Lorazepam; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Benadryl® Ativan® Decadron® (BAD) Pump (Experimental): Patients receive ondansetron hydrochloride IV twice daily and saline IV twice daily beginning 30-60 minutes prior to the start of chemotherapy. Patients also receive diphenhydramine hydrochloride, lorazepam, and dexamethasone by continuous infusion pump.
  Interventions: Drug: Decadron®; Drug: Benadryl®; Drug: Ativan®; Drug: ondansetron hydrochloride
- Control Arm Saline (Active Comparator): Patients receive ondansetron hydrochloride IV twice daily and dexamethasone IV twice daily beginning 30-60 minutes prior to the start of chemotherapy. Patients also receive saline by continuous infusion pump.
  Interventions: Drug: Decadron®; Drug: ondansetron hydrochloride

INTERVENTIONS:
Drug: Decadron® — Given IV
  Other Names: dexamethasone
Drug: Benadryl® — Given IV
  Other Names: diphenhydramine hydrochloride
  Arms: Benadryl® Ativan® Decadron® (BAD) Pump
Drug: Ativan® — Given IV
  Other Names: lorazepam
  Arms: Benadryl® Ativan® Decadron® (BAD) Pump
Drug: ondansetron hydrochloride — Given IV
  Other Names: Zofran; Ondisolv

SUMMARY:
RATIONALE: Diphenhydramine, lorazepam, and dexamethasone may help lessen or prevent nausea and vomiting in patients treated with chemotherapy. It is not yet known whether diphenhydramine, lorazepam, and dexamethasone are more effective than standard therapy in treating nausea and vomiting caused by chemotherapy.

PURPOSE: This randomized phase II trial is studying diphenhydramine, lorazepam, and dexamethasone to see how well they work compared with standard therapy in treating nausea and vomiting caused by chemotherapy in young patients with newly diagnosed cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the degree of chemotherapy-induced nausea and vomiting (CINV) in pediatric patients with newly diagnosed cancer treated with diphenhydramine hydrochloride, lorazepam, and dexamethasone vs standard antiemetic therapy during the first course of emetogenic chemotherapy.

Secondary

* Compare the degree of CINV during the first 3 days after completion of the first course of emetogenic chemotherapy in patients treated with these antiemetic regimens.

OUTLINE: This is a randomized, prospective, double-blind, multicenter study. Patients are stratified according to the emetogenic potential of their chemotherapy regimen (high vs moderate). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive ondansetron hydrochloride IV twice daily and saline IV twice daily beginning 30-60 minutes prior to the start of chemotherapy. Patients also receive diphenhydramine hydrochloride, lorazepam, and dexamethasone by continuous infusion pump.
* Arm II: Patients receive ondansetron hydrochloride IV twice daily and dexamethasone IV twice daily beginning 30-60 minutes prior to the start of chemotherapy. Patients also receive saline by continuous infusion pump.

In both arms, treatment continues during the first course of chemotherapy. Patients may also receive rescue antiemetic medication to control breakthrough nausea or emesis.

Patients and their parents complete the Adapted Rhodes Index of Nausea, Vomiting, and Retching- Measured by Child/Parent questionnaire once before beginning chemotherapy, twice daily during chemotherapy, and for 3 days after completion of chemotherapy.

PROJECTED ACCRUAL: A total of 180 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* ≥ 8 years of age and < 19 years of age at the time of registration
* Newly diagnosed with cancer
* Chemotherapy naive
* Scheduled to receive moderately or highly emetogenic chemotherapy (non-steroid containing regimen) as an in-patient. (Refer to Appendix IV. In multiple agent regimens, select the agent with the highest emetic potential.)
* Scheduled for placement of IV accesses device(s) for treatment purposes (allowing a dedicated line for continuous infusion of study agent)
* Not pregnant or lactating

EXCLUSION CRITERIA:

* Prior chemotherapy
* Central Nervous System disease
* Stem cell transplant while on-study
* Out-patient chemotherapy
* Steroids are included in their chemotherapy regimen
* Contraindication to the use of dexamethasone (e.g. diabetes)
* Hepatic and/or renal failure
* Allergic to any of the study medications
* Pregnant or lactating

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haydar Frangoul, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (7):
- United States (6):
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - St. Joseph's Children's Hospital of Tampa, Tampa, Florida
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - CHRISTUS Santa Rosa Children's Hospital, San Antonio, Texas
- San Jorge Children's Hospital, Santurce, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at participating SunCoast CCOP Research Base affiliated CCOPs and MB-CCOP institutions. Potential subjects may be provided with a paper study brochure that included a brief study overview by study staff. No recruitment or dissemination of any study brochures or materials occured prior to each site obtaining IRB approval.
Period: Overall Study
Arm/Group | Benadryl® Ativan® Decadron® (BAD) Pump | Control Arm Saline
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline number of participants was determined by the number of participants that completed their Baseline Study visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Benadryl® Ativan® Decadron® (BAD) Pump | Control Arm Saline | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 4 | 6
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Requiring Rescue Medication for Breakthrough Nausea or Emesis During Inpatient Chemotherapy
Description: Rescue medication is any medication administered by the treating team to control breakthrough nausea or emesis. Rescue medications were used to treat any patient who has enough symptoms requiring additional therapy. All patients were instructed to first use the push button on the pump. On-demand administration of study agent via the patient-controlled infusion pump will not be considered rescue therapy - it is part of the antiemetic treatment regimen. If on-demand administration is not successful in controlling the patient's symptoms, then as-needed rescue medications are to be administered. The treating staff will administer additional (as needed) doses of intravenous antiemetics, depending on the institutional preference.
Time Frame: during in-patient cycle of chemotherapy, up to 4 days
Measure: Number; unit: participants
Arm/Group | Benadryl® Ativan® Decadron® (BAD) Pump | Control Arm Saline
Number analyzed (Participants) | 3 | 4
participants | 1 | 3

2. Secondary Outcome: Proportion of Patients Requiring Rescue Medication for Breakthrough Nausea or Emesis After Completion of the First Course of Emetogenic Chemotherapy
Description: CINV will be determined based on the number of rescue medications used during the 3 days following completion of chemotherapy cycle. Rescue medication is any medication administered by the treating team to control breakthrough nausea or emesis. Rescue medications were used to treat any patient who has enough symptoms requiring additional therapy. All patients were instructed to first use the push button on the pump. On-demand administration of study agent via the patient-controlled infusion pump will not be considered rescue therapy - it is part of the antiemetic treatment regimen. If on-demand administration is not successful in controlling the patient's symptoms, then as-needed rescue medications are to be administered. The treating staff will administer additional (as needed) doses of intravenous antiemetics, depending on the institutional preference.
Time Frame: 3 days of following completion of first chemotherapy cycle
Measure: Number; unit: participants
Arm/Group | Benadryl® Ativan® Decadron® (BAD) Pump | Control Arm Saline
Number analyzed (Participants) | 3 | 4
participants | 3 | 4

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed daily beginning with the first cycle of chemotherapy and administration of study agent/placebo until 3 days following completion of chemotherapy cycle.
Description: AEs were assessed by study staff during in-patient chemotherapy, at discharge and 3 days following completion of chemotherapy with patient and patient's primary caregiver. AEs were also assessed using the Adapted Rhodes Index of Nausea, Vomiting and Retching Measured by Children and Parents that were completed twice daily.
Arm/Group | Benadryl® Ativan® Decadron® (BAD) Pump | Control Arm Saline
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benadryl® Ativan® Decadron® (BAD) Pump (N=3) | Control Arm Saline (N=4)
Pain associated with biopsy (Surgical and medical procedures) | 0 (0) | 1 (1) — Pain associated with biopsy required during in-patient chemotherapy. Biopsy not related to study treatment or procedures and was scheduled prior to subject going on study.

LIMITATIONS AND CAVEATS:
The study was closed prior to completing enrollment based on the recommendation by the SunCoast CCOP Research Base Data Safety Monitoring Board for a lack of feasibility and poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes